CLINICAL TRIAL: NCT03256487
Title: Intravenous Buprenorphine Versus Morphine for Severe Pain in the Emergency Department
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alameda Health System (Other)
Responsible Party: Principal Investigator, David Duong, Principal Investigator, Alameda Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB17-04172B
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Buprenorphine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The provider, nurse administering the medication, patient, and research assistant will be masked to the randomization and the drug provided. We will ensure masking by the following mechanisms: drugs will be prepared by the pharmacy staff in identical 10mL syringes; the medication will be diluted to a volume of 10mL with normal saline (NS); and both medications are clear so the syringes will appear identical. Both drugs will be administered over the same period of time, 3-5 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Buprenorphine (Experimental): Patients will receive IV buprenorphine 0.3mg diluted to a volume of 10mL with NS in a plastic syringe administered over 3-5 minutes. At 20 minutes, the patient will be asked "would you like more pain medication?" If he/she answers "yes", then he/she will receive a second dose of IV buprenorphine 0.3mg.
  Interventions: Drug: Buprenorphine
- Morphine (Active Comparator): Patients will receive IV morphine 0.1mg/kg (max dose 8mg) diluted to a volume of 10mL with NS in a plastic syringe administered over 3-5 minutes. At 20 minutes, the patient will be asked "would you like more pain medication?" If he/she answers "yes", then he/she will receive a second dose of IV morphine 0.1mg/kg (max dose 8mg).
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Buprenorphine — buprenorphine 0.3mg IV
  Arms: Buprenorphine
Drug: Morphine Sulfate — morphine 0.1 mg/kg IV (max 8mg per dose)
  Arms: Morphine

SUMMARY:
This study evaluates intravenous (IV) buprenorphine versus IV morphine for the management of severe, acute pain among emergency department (ED) patients. ED patients with severe pain will be randomized in equal proportion to receive IV buprenorphine or IV morphine.

DETAILED DESCRIPTION:
Buprenorphine is classified as a partial mu opioid agonist and a weak kappa antagonist. In lower doses, buprenorphine has an analgesic potency 25 to 40 times more potent than similar milligram dosages of morphine. Consistent with its partial agonist activity, an apparent ceiling effect for opioid-induced ventilatory impairment has been demonstrated. These properties would suggest that buprenorphine is an effective analgesic with a favorable safety profile.

Objective: The objective of this study is to determine if there is a clinically significant difference in reduction of pain scores, measured by the Numeric Rating Scale (NRS), between intravenous (IV) buprenorphine and IV morphine for severe pain in patients presenting to the Alameda Health System--Highland Hospital ED. The investigators are evaluating if IV buprenorphine is non-inferior to IV morphing. The investigators hypothesize that buprenorphine will provide equivalent analgesic effects as morphine at 60 minutes, with a lower proportion of medication adverse effects.

Study Design: This is a double-blinded, randomized controlled non-inferiority trial comparing the analgesic efficacy of intravenous buprenorphine versus intravenous morphine for ED patients presenting with severe, acute pain.

Participants: ED patients aged ≥18 years old who present with severe (pain NRS ≥7), acute pain warranting (according the treating provider's judgment) and able to receive IV opioid analgesia. The investigators will exclude pregnant patients, patients deemed too critically ill by the provider, patients with allergy to buprenorphine or morphine, patients in custody, patients on methadone, patients who have taken/received short acting opioid medications in the last 12 hours, and patients who have taken/received long acting opioid medication in the past 24 hours.

Intervention: In arm A, patients will receive IV Buprenorphine 0.3mg diluted to a volume of 10mL with NS in a plastic syringe administered over 3-5 minute. In arm B, patients will receive IV morphine 0.1mg/kg (max 10mg) over 3-5 minutes. In both arms, at 20 minutes the patient will be asked "would you like more pain medication?" If he/she answers "yes", then he/she will receive a second dose of the same amount of medication they previously received based on the randomized arm they were placed into. At the end of the study time, 60 minutes, the patient's ongoing pain management will be left to the attending physician caring for the patient in the ED.

Data Collection: For both arms, the patients' NRS pain scores and adverse effects will be queried at times 0, 10min, 20 min, 30min, 40min, 50 min, and 60 min. Demographic and comorbidity data points will be abstracted during or after the study's conclusion.

ELIGIBILITY:
Inclusion Criteria:

* ED patients with acute pain NRS ≥7 warranting IV opioid analgesia (according to ED provider)

Exclusion Criteria:

* Patient refusal
* pregnancy

  * level 1 trauma patients
  * patients deemed critically ill by provider
  * patients in custody
  * patients on methadone
  * Patients who have received or taken any short acting opioid medication in the past 12 hours.
  * Patients who have received or taken any long acting opioid medication in the past 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain score difference at 60 minutes | 60 minutes
  The difference in pain scores (measured by NRS) between the two arms at 60 minutes.

SECONDARY OUTCOMES:
Pain score difference at 50 minutes | 50 minutes
  The difference in pain scores (measured by NRS) between the two arms.
Pain score difference at 40 minutes | 40 minutes
  The difference in pain scores (measured by NRS) between the two arms.
Pain score difference at 30 minutes | 30 minutes
  The difference in pain scores (measured by NRS) between the two arms.
Pain score difference at 20 minutes | 20 minutes
  The difference in pain scores (measured by NRS) between the two arms.
Pain score difference at 10 minutes | 10 minutes
  The difference in pain scores (measured by NRS) between the two arms.
Adverse events | 10, 20, 30, 40, 50, and 60 minutes
  Hypertension (SBP > 180) from documented vital signs,hypotension (SBP <90) from documented vital signs, hypoxia (oxygen saturation < 90%), respiratory depression (RR<8 or need for mechanical intervention), nausea, vomiting, symptoms of opiate withdrawal (diarrhea, abdominal pain, diaphoresis)
Pain reduction | 10, 20, 30, 40, 50, and 60 minutes
  Pain reduction at each time point. Measured by NRS (time 0) minus NRS (time x)
Successful analgesia | 60 minutes
  Proportion of patients with NRS < 3 at 60 minutes
Repeat dosing | 20 minutes
  Proportion of patients requiring reducing of analgesia at 20 minutes
Summed Pain Intensity difference | 60 minutes
  Measurement combining relief magnitude and duration in a single score

CONTACTS AND LOCATIONS:
Locations (1):
- Alameda Health System, Highland Hospital, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No